CLINICAL TRIAL: NCT03078660
Title: Pilot Trial to Test a Nutrition Application for Making Smart and Healthy Choices When Purchasing Food in Grocery Stores
Brief Title: Pilot Trial to Test a Nutrition Application for Making Smart and Healthy Choices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A4540515
Record Dates: First submitted 2017-03-07; First posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Diet Modification; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Application (Experimental): Participants will have access to a smartphone application that provides a healthy shopping list based on requirements, budget and discounts to improve dietary practices and weight
  Interventions: Behavioral: Smartphone Application
- Traditional Nutritional Counseling (Active Comparator): Participants will participant in a face-to-face counseling session with a registered dietitian.
  Interventions: Behavioral: Traditional Nutritional Counseling

INTERVENTIONS:
Behavioral: Smartphone Application — The smartphone Application generates a shopping list for participants, based on a low caloric diet (energy requirements minus 500 kcals), taking into consideration the Dietary Guidelines for Americans' recommendations and also considering the available budget for each shopping event and the weekly discounts from major supermarkets.
  Arms: Smartphone Application
Behavioral: Traditional Nutritional Counseling — Participants will have a face-to-face counseling session with a registered dietitian, who will provide recommendations for a low caloric diet (energy requirements minus 500 kcals) using the food group sheets from the Dietary Guidelines for Americans.
  Arms: Traditional Nutritional Counseling

SUMMARY:
An innovative nutritional application (App) entitled "MyNutriCart" was developed to create a list of foods and beverages to help individuals make smart and healthy choices when purchasing foods at grocery stores based on the Dietary Guidelines for Americans. This App was tested in a pilot trial to evaluate its feasibility, usability, and acceptability for making smart and healthy choices when purchasing food in grocery stores and test its effectiveness in improving food selection, dietary patterns, and weight status compared with the traditional nutritional counseling.

DETAILED DESCRIPTION:
An innovative nutritional application (App) entitled "MyNutriCart" was developed to create a list of foods and beverages to help individuals make smart and healthy choices when purchasing foods at grocery stores based on the Dietary Guidelines for Americans. A pilot randomized clinical trial was done to test the effectiveness of this App on food selection and purchase, dietary patterns, and weight loss during two months of intervention. We also assessed feasibility, usability, satisfaction and acceptability of the App. A total of 138 overweight and obese adults aged 21-45 years old who own a Smartphone were invited to participate in this study. Participants were randomized into two groups; (1) the intervention group used the App, which generated a healthy grocery list to use when purchasing foods in in the supermarket; (2) the control group had a traditional intervention with a nutritionist. To assess the impact of the intervention on dietary patterns, participants completed three 24-hour dietary recalls, a short food frequency questionnaire (FFQ) and provided grocery receipts at baseline and at the end of the study (8 weeks later). Weight and height were also performed before and after the intervention. Feasibility, usability, satisfaction, and acceptability of the nutrition App were assessed at the end of the study using a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* overweight/obese adults
* aged 21-45 years
* main household shopper (responsible for >50% of the household grocery shopping)
* shopping at a grocery store at least once a week
* owner of a smartphone (iPhone or Android) with internet access
* willingness to be randomized into one of the two groups.

Exclusion Criteria:

* Use of other apps
* Participating in weight loss programs
* Pregnant women
* Individuals with chronic health conditions
* Individuals with reported food allergies

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of food intake | 8 weeks
  A Food frequency questionnaire was completed by participants at baseline and end of study. It includes the frequency of consumption of the following food groups: fruits, vegetables, starchy vegetables, refined and whole grains, legumes, healthy proteins, red meats, cold cuts and cured meats, whole-fat and low-fat dairy products, 100% fruit juices, and sugar-sweetened beverages.
Change in food intake | 8 weeks
  Three 24-h recalls were completed by participants at baseline and end of study. The consumption of the following food groups was analyzed: fruits, vegetables, starchy vegetables, refined and whole grains, legumes, healthy proteins, red meats, cold cuts and cured meats, whole-fat and low-fat dairy products, 100% fruit juices, and sugar-sweetened beverages.
Change in foods selection | 8 weeks
  Grocery receipts were evaluated at baseline and end of study for changes in food purchase of the following food groups: fruits, vegetables, whole grains, 100% fruit juices, and sugar-sweetened beverages.

SECONDARY OUTCOMES:
Change in weight | 8 weeks
  Weight will be assessed at baseline and end of study
Feasibility | 8 weeks
  Participants completed a questionnaire with 3 questions about feasibility, in which they rated each item using a five point Liker scale ranging from strongly agree (5 points) to strongly disagree (1 point): (1) easiness to use the App; (2) easiness to learn how to use the App; and (3) easiness how to find information in the App.
Usability | 8 weeks
  Participants completed a questionnaire with 1 question about usability: times the App was used.
Satisfaction | 8 weeks
  Participants completed a questionnaire with 3 questions about their satisfaction with the App, in which they rated each item using a five point Liker scale ranging from strongly agree (5 points) to strongly disagree (1 point). These items were: (1) satisfaction with information provided; (2) likenesses of re-using the app; (3) overall likeness and rating of the App.
Acceptability | 8 weeks
  Participants completed a questionnaire with 3 questions about the acceptability of the App, in which they rated each item using a five point Liker scale ranging from strongly agree (5 points) to strongly disagree (1 point). These items were: (1) attractiveness of the App; (2) comfortable using the app; (3) overall likeness about the layout and screen of the App.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Palacios, PhD, Principal Investigator — Nutrition Program, School of Public Health, Medical Sciences Campus, University of Puerto Rico
Locations (1):
- University of Puerto Rico, Medical Sciences Campus (UPR-MSC), San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
No plan yet